CLINICAL TRIAL: NCT02386228
Title: miRNA Markers of Hydrocephalus in Intraventricular Hemorrhage (IVH)
Brief Title: Micro Ribonucleic Acid (miRNA) Markers of Hydrocephalus in Intraventricular Hemorrhage (IVH)
Status: Terminated | Type: Observational
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Translational Genomics Research Institute (Other)
Responsible Party: Principal Investigator, Madelon Petersen, Research Clinician, St. Joseph's Hospital and Medical Center, Phoenix
Other Study IDs: 14BN104
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Intraventricular Hemorrhage; Spina Bifida
Keywords: miRNA; posthemorrhagic hydrocephalus (PHH)
MeSH Terms: conditions — Spinal Dysraphism | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CSF and blood
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: collection of CSF and blood — collection of CSF and blood

SUMMARY:
A collection of biological samples (cerebrospinal fluid [CSF] and blood) from patients under 6 years of age who are diagnosed with intraventricular hemorrhage or spina bifida.

DETAILED DESCRIPTION:
IVH is an important cause of brain injury in newborns and more so in those born prematurely. Depending on the severity of the hemorrhage and the care provided the newborn, the impact of IVH can range from a temporary issue with no permanent consequences to a life-threatening condition with severe neurodevelopmental sequelae. The outcomes of patients with IVH are not only dictated by the direct effects of the hemorrhage, but to associated processes such as hydrocephalus, periventricular infarction and leukomalacia. Despite the availability of better diagnostic and therapeutic tools, the incidence of IVH has remained constant over the past 50 years, and is mostly due to the increased survival rates of very low weight premature infants. Recent statistics demonstrate that close to 12,000 premature infants develop IVH in the United 'states every year and more than 50% of them develop some degree of posthemorrhagic hydrocephalus (PHH). It is believed that PHH originates as a result or arachnoiditis, gliosis, and subsequent fibrosis impairing the flow and reabsorption of cerebrospinal fluid (CSF). Despite the lack of clarity about the pathogenesis of PHH, it is well accepted that its presence exacerbates the damage caused by the hemorrhage to the periventricular white matter. Multiple efforts have been made to identify the mechanisms and mediators of the development of PHH and white matter damage. Molecules such as transforming growth factor-beta (TGF-beta) have been demonstrated to enhance the expression of genes encoding for fibronectin, collagen and other extracellular matrix components. Unfortunately, not enough evidence has been generated to be able to envision a potential solution for the problem. The current management of PHH is focused on controlling the damage that pressure, distortion, and/or ischemia may cause to the immature brain. Direct evacuation of ventricular contents with CSF diversion mechanisms remains, such as sequential lumber punctures, external ventricular draining, and reservoir placement. Intraventricular fibrinolytic therapy or permanent shunting represent most effective tools by mechanically evacuating bleeding products and preventing the accumulation of CSF. However, they are all highly invasive techniques that carry major risks and complications. The use of diuretics has been presented as a non-invasive alternative, but the results prove them inefficient. Extracellular miRNA sequences have been found to be major modulators of protein coding genes involved in differentiation, proliferation, and apoptosis. Several studies have reported the presence of significant amounts of miRNA in extracellular fluids such as plasma, urine, saliva, and semen. The researchers believe that extracellular miRNAs are present in CSF and that sequential evaluation of their expression can provide a unique biomarker signature, time sensitive enough to reflect the evolution of pathological events underlying the development of PHH. The identification of a miRNA biomarker for PHH development and/or hemorrhagic related injury would also be a means to quickly evaluate treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Age between 0 and 6 years.
* Diagnosis of IVH or spina bifida
* Granted access to CSF and blood via surgery, CSF diversion device, venous access, and/or arterial access.

Exclusion Criteria:

* Older than 6 years.
* Diagnosis of infection or other acute inflammatory process involving the central nervous system.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants with IVH or spina bifida
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
miRNA sequences | within 30 days of blood or CSF collection
  Identification of miRNA sequences common to patients with IVH and patients with spina bifida to determine condition specific expression profiles, multivariate analysis of candidate miRNA sequences that are differentially expressed between the two conditions but between different outcomes (development of hydrocephalus) to target potential markers. Once identified, mechanisms for the rapid detection of marker sequences will be developed and their predictive value tested in future collections.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Spetzler, MD, Principal Investigator — Barrow Brain and Spine physician with SJHMC privileges
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States